CLINICAL TRIAL: NCT02572661
Title: Mapping of Sentinel Lymph Node Drainage Using SPECT to Tailor Highly-Selective Elective Nodal Irradiation in Node-Negative Neck of Patients With Head and Neck Cancer (SUSPECT)
Brief Title: Mapping of Sentinel Lymph Node Drainage Using SPECT (SUSPECT) (SUSPECT)
Acronym: SUSPECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N14SUS; N14SUS (Registry Identifier: PTC); NL51706.031.14 (Registry Identifier: CCMO)
Record Dates: First submitted 2014-12-22; First posted 2015-10-09 (Estimated); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Head and Neck Cancer
Keywords: Radiotherapy, Sentinel Node Mapping, Spect
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Squamous Head and Neck Cancer (Other): radiation
  Interventions: Radiation: radiation in Squamous Head and Neck Cancer

INTERVENTIONS:
Radiation: radiation in Squamous Head and Neck Cancer

SUMMARY:
This study aims to explore the feasibility, safety and outcome of a non-invasive sentinel node mapping (SNM) to individually tailor the elective nodal irradiation (ENI) to the ipsilateral neck only and to exclude the contralateral negative neck from the irradiation fields when there is no draining sentinel node. Subsequently the dose to the salivary glands, mucosal area and the swallowing and chewing muscles and structures involved in voicing and articulation will significantly be reduced

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with histopathologic proven primary HNSCC (T1 -3 N0 -1) located in the oral cavity, oropharynx, larynx (except T1 glottic ), and hypopharynx, not crossing the midline and planned for treatment with (chemo)radiotherapy in curative setting
* No chemotherapy or surgery prior to inclusion
* No distant metastatic spread at the time of inclusion
* Age ≥ 18 years
* WHO performance status 0 or 1
* Signed written informed consent

Exclusion Criteria:

* Patients with previously radiation treatment in the head and neck region, for any reason
* Patients with previous neck dissection
* Patients with recurrent or second primary tumor in the head and neck region
* Patients with head and neck malignancies arising from skin, lip, nose, sinuses, nasopharynx, salivary glands, thyroid gland or esophagus
* Previous history of cancer in the last five years (excluding basal cell carcinoma of the skin and in situ SCC of the cervix)
* Pregnancy or no active contraception for pre-menopausal women
* Known hypersensitivity to iodine or nanocolloid injection
* Having any condition (physical, mental, sociological) that interferes with the informed consent procedure and follow up schedules

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-07-23 (Actual); Primary Completion 2018-11-09 (Actual); Study Completion 2018-11-09 (Actual)

PRIMARY OUTCOMES:
Feasibility and safety of single side radiation therapy measured by physical examination and toxicity measurement by CTCAE 4.03 at 12 weeks | 12 weeks
  mapping of sentinel lymph node drainage to indentify groups at low risk of the probability of contra regionale failure is to be estimated to be 2% at 2 years. A recurrrence rate of >15% will be assumed unacceptable

CONTACTS AND LOCATIONS:
Overall Officials: Abrahim Al-Mamgani, MD, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- the Netherlands Cancer Instiute, Amsterdam, Netherlands